CLINICAL TRIAL: NCT00596011
Title: Phase II, Randomized, Double-blind, Multi-centered Study of Polyphenon E in Men With High-grade Prostatic Intraepithelial Neoplasia (HGPIN) or Atypical Small Acinar Proliferation (ASAP)
Brief Title: Study of Polyphenon E in Men With High-grade Prostatic Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCC-15008; R01CA12060-01A1 (Other: NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Prostatic Hyperplasia
Keywords: prostate cancer; PIN; polyphenon E; EGCG
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyphenon E Treatment (Active Comparator): Polyphenon E, 200 mg epigallocatechin gallate (EGCG) twice a day (BID)
  Interventions: Drug: Polyphenon E
- Placebo Administration (Placebo Comparator): Matching placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyphenon E — Polyphenon E, at a dose of 400 mgs EGCG (200 mgs BID) for 1 year in men diagnosed with HGPIN and ASAP.
  Other Names: green tea catechins; PolyE
  Arms: Polyphenon E Treatment
Drug: Placebo — Matching placebo BID
  Arms: Placebo Administration

SUMMARY:
The purpose of this study was to determine whether the daily consumption of decaffeinated green tea catechins (Polyphenon E®) for 1 year reduces the rate of progression to prostate cancer (PCa) in men diagnosed with HGPIN or ASAP. The aim was to recruit and treat 240 (120 men/arm) men diagnosed with the prostate condition HGPIN or ASAP with a capsule form of standardized green tea extract called Polyphenon E or placebo for a 12-month period and see if it can prevent progression of the prostate condition to prostate cancer. Investigators wanted to see if Polyphenon E reduces lower urinary tract symptoms and if this can be taken safely over one year. Investigators wanted to study how Polyphenon E is able to slow the progression to prostate cancer, or the mechanism of action of Polyphenon E. If the safety and the effects of Polyphenon E on slowing down the progression of prostate cancer is shown in our study, this will be a safe way of treating men who are at high risk or men like you who have a prostate condition that increases your chances of getting prostate cancer, so that we can prevent prostate cancer in the future.

DETAILED DESCRIPTION:
At the baseline/randomization visit, a QOL (Medical Outcomes Study Short Form-36) and lower urinary tract symptoms (LUTS) score assessment will be completed; urine and serum will be collected for measurement of diagnostic markers; plasma will be collected for measurement of baseline catechin levels; serum will be collected for banking; and diet recall forms will be collected. Participants will be equally randomized to blinded treatment with either Polyphenon E 200 mg EGCG bid or matching placebo, and an initial supply of study drug will be dispensed. All participants will also be provided with a standard multivitamin/mineral supplement to assure consistent, appropriate nutrient intake among study participants. The planned intervention period is 12 months; participants will return for monthly clinic visits during the intervention period. At each monthly clinic visit, blood will be drawn for repeat hepatic function panel, lactate dehydrogenase (LDH) and prothrombin time/partial thromboplastin time (PT/PTT), and participants will be interviewed to review and capture information from study agent intake log (pill count), assess signs and symptoms and concomitant medications; additional study medication will be dispensed as needed. After 3 and 6 months of intervention, blood will be drawn for serum chemistry and hematology, and LUTS and QOL assessments will be performed. In addition, at the 6 month visit, two-day diet recall forms will be collected, blood will be drawn for plasma catechin measurements and serum banking, serum and urine will be collected for diagnostic marker measurement, and repeat digital rectal exam (DRE) and prostate specific antigen (PSA) will be performed. If there is a palpable prostate nodule or confirmed PSA increase (>0.75 ng/ml) at 6 months, a repeat biopsy will be performed. If the 6-month biopsy shows evidence of disease progression, participants will stop intervention and proceed to the post-intervention assessment; otherwise, intervention will continue through month 12. At the end of intervention (maximum of 12 months), a repeat prostate biopsy will be performed for post-intervention endpoint measurements. In addition, the physical exam and DRE, LUTS and QOL will be repeated, and 2-day diet recall forms will be collected. Blood will be drawn for serum chemistry and hematology, PSA, hepatic function panel, LDH, PT/PTT; serum and urine will be collected for diagnostic marker measurement; plasma will be collected for catechin measurements; and serum will be collected for banking. Participants will be interviewed to review and capture information from study agent intake log (pill count), assess signs and symptoms and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Men with a diagnosis of HGPIN or ASAP in a minimum of 1 of 8 cores from a biopsy performed within six months of study entry. Diagnosis of HGPIN or ASAP (which includes men with ASAP and HGPIN) via trans-rectal ultrasound (TRUS biopsy) is also considered acceptable for inclusion.
* Prostate biopsy with a minimum of 8 cores performed within 6 months of study entry that shows no evidence of cancer.
* 30-80 years of age at the time of registration
* PSA ≤10 ng/ml
* Omnivorous diet
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Participants must have normal organ and marrow function as demonstrated by the following parameters being within normal institutional limits: complete blood count (CBC); liver function tests (LFTs); albumin, total and direct bilirubin, alkaline phosphatase, aspartic transaminase (AST), alanine transaminase (ALT), and total protein), PT/PTT, and LDH; serum creatinine <1.5 mg/dl or measured creatinine clearance 60 cc/min
* Absence of consumption of toremifene citrate, finasteride, testosterone, dehydroepiandrosterone (DHEA) or other testosterone-like supplements or medications which have known impact on PSA within 30 days of informed consent, or dutasteride within 90 days of informed consent
* Absence of consumption of any nutritional or herbal supplements containing green tea or green tea polyphenols
* No or low regular tea consumption (no more than 3 servings of hot tea or 6 servings of iced tea per week)
* Willing to discontinue current vitamin/mineral supplement use and substitute with a standard multivitamin supplement provided for the study
* Willing to use an effective method of contraception, if the partner is of child-bearing age, while on study
* Willing to comply with proposed visit and treatment schedule
* Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Evidence of acute prostatitis or urinary tract infection at the time of PSA measurement; men may be enrolled 30 days after completion of treatment, provided all other eligibility criteria are met
* Current or prior history of prostate cancer or other malignancies (exceptions include non-melanoma skin cancer or other cancer with no evidence of tumor recurrence 5 years after definitive treatment)
* History of renal or hepatic disease, including history of hepatitis B, C or delta
* Participation in any other investigational study or use of any other investigational agents within 30 days of study entry
* History of allergic reactions attributed to tea or other compounds of similar chemical or biologic composition to Polyphenon E or the inactive components present in Polyphenon E and placebo capsules.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any psychological, familial, sociological or other concomitant condition that would not allow adequate compliance with the study protocol
* History of medical conditions that may predispose the participant to gastrointestinal bleeding (acute or chronic gastritis or colitis, or acute diverticulitis or hemorrhoids)
* Members of all races and ethnic groups are eligible for this trial. Since this is an investigation targeting men with HGPIN or ASAP, women are not eligible for the study.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, PhD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (10):
- United States (10):
  - University of Florida/Shands-Department of Urology, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Watson Clinic Center for Research, Inc., Lakeland, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - James A Haley VA, Tampa, Florida
  - University of Chicago - Department of Surgery, Chicago, Illinois
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Jefferson Medical College - Department of Urology, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Kim SJ, Amankwah E, Connors S, Park HY, Rincon M, Cornnell H, Chornokur G, Hashim AI, Choi J, Tsai YY, Engelman RW, Kumar N, Park JY. Safety and chemopreventive effect of Polyphenon E in preventing early and metastatic progression of prostate cancer in TRAMP mice. Cancer Prev Res (Phila). 2014 Apr;7(4):435-44. doi: 10.1158/1940-6207.CAPR-13-0427-T. Epub 2014 Feb 5. PMID 24501325
- [Result] Kumar NB, Pow-Sang JM, Spiess PE, Park JY, Chornokur G, Leone AR, Phelan CM. Chemoprevention in African American Men With Prostate Cancer. Cancer Control. 2016 Oct;23(4):415-423. doi: 10.1177/107327481602300413. PMID 27842331
- [Result] Kumar NB, Pow-Sang J, Spiess PE, Park J, Salup R, Williams CR, Parnes H, Schell MJ. Randomized, placebo-controlled trial evaluating the safety of one-year administration of green tea catechins. Oncotarget. 2016 Oct 25;7(43):70794-70802. doi: 10.18632/oncotarget.12222. PMID 28053292
- [Result] Kumar NB, Patel R, Pow-Sang J, Spiess PE, Salup R, Williams CR, Schell MJ. Long-term supplementation of decaffeinated green tea extract does not modify body weight or abdominal obesity in a randomized trial of men at high risk for prostate cancer. Oncotarget. 2017 Jun 29;8(58):99093-99103. doi: 10.18632/oncotarget.18858. eCollection 2017 Nov 17. PMID 29228755
- [Derived] Kumar NB, Pow-Sang J, Egan KM, Spiess PE, Dickinson S, Salup R, Helal M, McLarty J, Williams CR, Schreiber F, Parnes HL, Sebti S, Kazi A, Kang L, Quinn G, Smith T, Yue B, Diaz K, Chornokur G, Crocker T, Schell MJ. Randomized, Placebo-Controlled Trial of Green Tea Catechins for Prostate Cancer Prevention. Cancer Prev Res (Phila). 2015 Oct;8(10):879-87. doi: 10.1158/1940-6207.CAPR-14-0324. Epub 2015 Apr 14. PMID 25873370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the Moffitt Cancer Center and 7 other sites in the United States, from September 2008- March 2013.
Pre-assignment Details: Participants were block randomized by diagnosis to receive Polyphenon E®) (PolyE) containing 400 mgs (-)-epigallocatechin-3-gallate (EGCG) per day (n=49) or placebo (n=48) for 1 year.
Groups:
- Active Comparator: Polyphenon E Treatment: Polyphenon E, 200 mg epigallocatechin gallate (EGCG) twice a day (BID)
- Placebo Comparator: Placebo Administration: Matching placebo twice a day (BID)
Period: Overall Study
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Started | 49 | 48
Completed | 36 | 38
Not Completed | 13 | 10
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 11 | 7

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Full Range); unit: years] | 62 [45 to 79] | 64.10 [45 to 78] | 63.02 [45 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 22 | 23 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 49 | 48 | 97
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression to Prostate Cancer (PCa)
Description: Number of participants with diagnosis of high-grade prostatic intraepithelial neoplasia (HGPIN) or atypical small acinar proliferation (ASAP) who progressed to prostate cancer (PCa) at one year.
Time Frame: 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 49 | 48
participants | 4 | 6

2. Primary Outcome: Rate of Progression From HGPIN to ASAP or PCa
Description: Analyses of participants reaching a definitive endpoint. Number of baseline HGPIN participants who progressed to ASAP or PCa.
Time Frame: 12 months
Population: Baseline HGPIN participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 26 | 25
participants
  Progressed to ASAP or PCa | 3 | 10
  Progressed to ASAP | 0 | 5

3. Secondary Outcome: Treatment Emergent Adverse Events (AEs)
Description: Safety of Polyphenon E (200 mg EGCG bid for one year) in men with HGPIN or ASAP. Number of participants with AEs Possibly or Probably related to treatment.
Time Frame: 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 49 | 48
participants
  Definitely related to treatment | 0 | 0
  Probably related to treatment | 5 | 1
  Possibly related to treatment | 7 | 3
  Unlikely to be related to treatment | 7 | 9
  Unrelated to treatment | 193 | 156
  Total | 212 | 169

4. Secondary Outcome: Occurrence of Grade 3 or Higher Adverse Events (AEs)
Description: Number of participants with AEs grade 3 or higher, per treatment arm.
Time Frame: 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 49 | 48
participants | 10 | 3

5. Secondary Outcome: Median Serum Total Prostatic Specific Antigen (tPSA)
Description: Median ng/mL serum tPSA post treatment, per treatment arm.
Time Frame: 12 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 49 | 48
ng/mL | 3.5 [2.80 to 5.10] | 4.90 [3.65 to 6.15]

6. Other Pre Specified Outcome: Change in Scores - Lower Urinary Tract Symptom (LUTS)
Description: Change in score from baseline to 1 year. LUTS represent a common conglomeration of storage, voiding, and post-micturition symptoms with reported debilitating effect on quality of life. Symptom severity related to urinary frequency, nocturia, weak urinary stream, hesitancy, intermittency, incomplete bladder emptying and urinary urgency are assessed. We utilized the American Urological Association Symptom Score for the evaluation LUTS in this patient population. Symptom Frequency Scores: 0 = Not at all, 1 = Less than 1 time in 5, 2 = Less than half the time, 3 = About half the time, 4 = More than half the time, 5 = Almost always. Total Symptom Score = Sum of individual scores of the 7 symptoms. (minimum possible score=0; maximum possible score =35; Range of scores and significance: 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms.
Time Frame: 1 year
Population: Participants with LUTS symptom scores available at baseline and at one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Number analyzed (Participants) | 29 | 28
units on a scale
  Incomplete empty - change | 0.07 (1.77) | 0.39 (1.99)
  Frequent urination - change | 0.03 (1.61) | 0.50 (1.45)
  Intermittency - change | 0.21 (1.32) | -0.04 (1.4)
  Nocturia - change | 0.31 (1.42) | 0.25 (1.69)
  Straining - change | 0.24 (0.99) | 0.25 (0.97)
  Urgency - change | 0.10 (1.47) | -0.25 (1.86)
  Weak stream | 0.24 (1.12) | 0.15 (1.49)
  Total Symptom Score - change | 1.21 (6.56) | 1.36 (7.93)

7. Other Pre Specified Outcome: Effect of Polyphenon E on the Fundamental Molecular Pathways
Description: Explore the effects of Polyphenon E on the fundamental molecular pathways contributing to chemopreventive activity of Polyphenon E in the prostate. This exploratory aim is ongoing.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Average of 12 months
Description: All participants. All adverse events, regardless of causality.
Arm/Group | Active Comparator: Polyphenon E Treatment | Placebo Comparator: Placebo Administration
Serious Adverse Events (participants affected / at risk) | 4/49 | 2/48
Other Adverse Events (participants affected / at risk) | 47/49 | 44/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Polyphenon E Treatment (N=49) | Placebo Comparator: Placebo Administration (N=48)
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac General - Other - Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term - Death NOS (General disorders) | 1 (1) | 0 (0)
Perforation, GI - Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection with unknown ANC - Wound (Infections and infestations) | 1 (1) | 0 (0)
Obstruction, GU - Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Polyphenon E Treatment (N=49) | Placebo Comparator: Placebo Administration (N=48)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 23 (53) | 26 (61)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 (14) | 8 (8)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 8 (8) | 9 (9)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 7 (10) | 6 (8)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (8) | 3 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (8) | 2 (7)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Creatinine (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 11 (20) | 16 (26)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Gastrointestinal - Other (Gastrointestinal disorders) | 7 (9) | 5 (8)
Nausea (Gastrointestinal disorders) | 6 (8) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (4) | 1 (1)
Pain - Head/headache (General disorders) | 10 (13) | 2 (8)
Pain - Extremity-limb (General disorders) | 3 (5) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 8 (11) | 10 (14)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3) | 3 (3)
Constitutional Symptoms - Other (General disorders) | 4 (4) | 7 (11)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3) | 2 (2)
Coagulation - Other (Investigations) | 7 (13) | 3 (8)
PTT (Partial Thromboplastin Time) (Investigations) | 5 (6) | 2 (2)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 4 (6) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 8 (11) | 2 (2)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Primary Endpoint: Progression to PCa. Recent evidence demonstrates ASAP is a stronger diagnostic predictor associated with PCa compared to HGPIN. Due to this evidence and recruitment challenges, we revised inclusion criteria to include men with ASAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes